CLINICAL TRIAL: NCT05336305
Title: Effects of Polydextrose Supplementation on Constipation in Patients Undergoing Hemodialysis
Brief Title: Polydextrose for Patients With Chronic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal Fluminense (Other)
Responsible Party: Principal Investigator, Denise Mafra, professor, Universidade Federal Fluminense
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DeniseMafra15
Record Dates: First submitted 2022-03-06; First posted 2022-04-20 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Chronic Kidney Diseases; Constipation
MeSH Terms: conditions — Renal Insufficiency, Chronic; Constipation | interventions — polydextrose

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Group (Placebo Comparator): Administration of corn starch daily for 2 months
  Interventions: Dietary Supplement: Polydextrose
- polydextrose (Experimental): Administration of 12g polydextrose daily for 2 months
  Interventions: Dietary Supplement: Polydextrose

INTERVENTIONS:
Dietary Supplement: Polydextrose — Administration of 3g polydextrose per day, for 2 months

SUMMARY:
Constipation is a common complication in patients with chronic kidney disease (CKD), especially in hemodialysis (HD) patients. Reduced intake of fibre-rich food is among the most important causes of constipation. The study aims to investigate the possible influence of polydextrose (PDX) supplementation on constipation in patients with CKD on HD.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Chronic Kidney Disease
* Hemodialysis patients for more than 6 months
* Aged 18 years or older

Exclusion Criteria:

* Patients pregnant
* Smokers
* Using antibiotics in the last 3 months
* Autoimmune diseases
* Clinical diagnosis of infectious diseases
* Clinical diagnosis of Cancer
* Clinical diagnosis of AIDS

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-03-30 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Change constipation status after supplementation with polydextrose | 2 months
  Stool frequency and Bristol Stool Form
Change in cytokines plasma levels measured by ELISA after supplementation with polydextrose | 2 months
  cytokines levels

CONTACTS AND LOCATIONS:
Locations (1):
- Denise Mafra, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Borges NA, Sahiun E, Ribeiro-Alves M, Regis B, Mafra D. Effects of Polydextrose Supplementation on Intestinal Function in Hemodialysis Patients: A Double-Blind, Randomized, Placebo-Controlled Trial. J Ren Nutr. 2023 Nov;33(6):747-754. doi: 10.1053/j.jrn.2023.06.008. Epub 2023 Jun 14. PMID 37321430